CLINICAL TRIAL: NCT05207098
Title: Pilot Study of Radiation-Associated Neurocognitive Function Among Head and Neck Cancer Patients
Brief Title: A Study of Neurocognitive Tests and Questionnaires for People With Head and Neck Cancer Who Are Undergoing Radiation Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-498
Record Dates: First submitted 2021-12-22; First posted 2022-01-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer
Keywords: Neurocognitive function; Neurocognitive Tests; Questionnaires; 21-498
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Mental Status and Dementia Tests; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurocognitive Tests and Questionnaires: The performance-based measures will be administered with a total completion time estimated to be 90 minutes. The neurocognitive battery is similar in content and duration to multiple previous and ongoing studies being conducted by the Neurocognitive Research Lab.
  Interventions: Other: Neurocognitive Tests; Other: Questionnaires

INTERVENTIONS:
Other: Neurocognitive Tests — Baseline only: WRAT Reading Test, WMS-IV Logical Memory Subtest, Hopkins Verbal Learning Test (HVLT), Oral Trailmaking - Part A and B, NAB Digit Span, Category Fluency Test, Oral Symbol Digit Modalities Test, Brief Test of Attention, FAS - Controlled Oral Word Association Test (COWAT), Verbal Naming, Enformia Cogsuite Battery
Other: Questionnaires — Sociodemographics, Computerized Cognitive Training Programs Questionnaire, CDC Behavioral Risk Factor (Smoking Assessment), Alcohol Consumption CDC, Current Health Rating (KPS), OARS Physical Health section, COVID Medical History, Hospital Anxiety and Depression Scale (HADS), Fatigue Symptom Inventory (FSI), Functional Assessment of Cancer Therapy-General (FACT-G V4), Functional Assessment of Cancer Therapy-Cognition (FACT-Cog V3), Sensory Gating Inventory (SGI)

SUMMARY:
The researchers are doing this study to collect more information about if, and how, neurocognitive function may be affected in people being treated with radiation therapy for head and neck cancer. Part of this study is to see if patients diagnosed with head and neck cancer who are undergoing radiation therapy are able to complete neurocognitive testing and questionnaires at 3 times over a period of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of a head and neck cancer, specifically these subtypes: nasopharynx, maxillary sinus, tonsil, base of the tongue, oral cavity, or larynx/hypopharynx, oropharynx, cancer of unknown primary, or salivary gland.
* Ages ≥ 18 and <89 at time of diagnosis.
* Recently diagnosed with their initial head and neck cancer and able to be consented prior to OR within first week of starting standard of care radiation therapy.
* Baseline simulation whole-brain MRI or CT available as part of standard of care.
* Patients diagnosed with cancer, no distant metastases.
* Karnofsky Performance Status of >= 70 or comparable ECOG performance at enrollment.
* As per self-report, if currently taking psychoactive medications (excluding gabapentin and including but not limited to antidepressants, and anxiolytics) on a daily basis, dose must have been stable for at least two months prior to enrollment.
* English fluent as per self-reported fluency of "well' or "very well", and having a reasonable comprehension of the study conversation in the opinion of the research staff).** ** Language verification: Prior to enrollment, all patients will be asked the following two questions by the CRC to verify English fluency necessary for participation in the study:

  1. How well do you speak English?

     Must respond "Well" or "Very well" when given the choices of:

     Very well, Well, Not well, Not at all, Don't know, or Refused.
  2. What is your preferred language for healthcare? Must respond English.

Exclusion Criteria:

* Patients with multiple primary head and neck cancers, carcinoma of unknown primary, or recurrence.
* Patients who previously received radiation therapy to the head and neck region as treatment for any prior cancer for any other non-cancerous condition.
* Patients who had chemotherapy within two years prior to their recent diagnosis of head and neck cancer, such as patients who received chemotherapy as treatment for any other type of cancer or received neoadjuvant chemotherapy prior to surgery to treat their recent head and neck diagnosis. Patients who receive induction chemotherapy just prior to the start of their radiation therapy or receive concurrent chemotherapy to treat their recent head and neck diagnosis are allowed
* At the discretion of the clinician, patients who are unable to comfortably speak due to symptoms of their cancer or treatment, such as surgery.
* Pre-existing diagnosis of neurodegenerative disorder that affects cognitive function (e.g. Alzheimer's disease, Parkinson's disease, Multiple Sclerosis, Dementia, Seizure Disorders, etc.).
* As per medical record or self-report, history of stroke or head injury requiring medical care, confirmed structural lesion on neuroimaging, and persistent cognitive difficulties impacting work or daily life or required cognitive rehabilitation.
* Pre-existing diagnosis of a Schizophrenia Spectrum Disorder, substance use disorder, Bipolar Disorder or Schizotypal personality disorder. Schizophrenia Spectrum Disorders include Schizophrenia, Schizophreniform disorder, Schizoaffective disorder, Delusional disorder, Brief psychotic disorder, and Attenuated Psychotic Disorder.
* Pre-existing visual or auditory impairment that would preclude ability to complete the assessments (e.g. history of significant macular degeneration or being unable to correct hearing with hearing aids)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSK patients at any location, diagnosed with HNC (nasopharynx, maxillary sinus, tonsil, base of the tongue, oral cavity, and larynx/hypopharynx).
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of newly diagnosed head and neck cancer patients recruited and retained on study | 1 year
  have complete the neurocognitive testing

CONTACTS AND LOCATIONS:
Overall Officials: Jonine Bernstein, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm